CLINICAL TRIAL: NCT02525354
Title: Obesity and Atopic-related Respiratory Disease: Possible Role of Dietary Omega 6 and 3 Fatty Acids
Brief Title: Dietary Arachidonic Acid, Obesity and Atopic Respiratory Disease
Status: Completed | Type: Observational
Sponsor: University of New Hampshire (Other)
Responsible Party: Principal Investigator, Anthony R. Tagliaferro, Professor of Human Nutrition, University of New Hampshire
Other Study IDs: UNH-01-2536-01
Record Dates: First submitted 2015-06-15; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Allergy; Obesity
Keywords: arachidonic aci; adiposity; atopy
MeSH Terms: conditions — Hypersensitivity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiological studies have shown obesity to be a risk factor of asthma. Research evidence of obesity and atopic(ie. allergic)-related respiratory diseases, has been less clear. The purpose of the present study was to test the hypothesis that the relationship between obesity and atopic-related respiratory disease in premenopausal women is mediated by a dietary imbalance of omega 6 and 3 polyunsaturated fatty acids.

DETAILED DESCRIPTION:
Sixty young adult obese and non obese women, with, and without asthma, were studied using a cross-sectional design. Body composition was measured by plethysmography. A fasted blood sample was taken to measure: specific and total immunoglobulin (IgE) antibodies,biochemical markers of atopy; glucose and insulin to measure insulin sensitivity; estrogen(17β-estradiol) and sex hormone-binding globulin to measure estrogen status of the women; hormone-products of fat tissue ( leptin, adiponectin, resistin, tumor necrosis factor alpha (TNFα), interleukins (IL-6,IL-18), that have been associated with both obesity and immune processes involved in asthma and allergy. Dietary intake of omega 6: linoleic acid (LA), arachidonic acid(AA); and omega 3 fatty acids: α linolenic (ALA), eicosapentanoic (EPA) and docosahexanoic (DHA) and other nutrients were assessed by food frequency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* For asthmatics, only individuals that were willing and capable of not using asthma medications for two days prior to laboratory testing.

Exclusion Criteria:

* An individual was excluded from the study if she had a history of high blood pressure, diabetes, heart disease, cigarette smoking, or eating disorders.
* Women that were pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female subjects were recruited from the University and surrounding local communities, using posted flyers, website announcements, personal announcements in classes, referrals from local physicians, and word of mouth. Prospective subjects were interviewed initially by telephone.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2001-10; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Predictors of serum concentration of specific and total IgE antibodies in obesity | one day
  Measures of insulin sensitivity, plasma concentrations of leptin, adiponectin, , estrogen, IL-18,and dietary arachidonic, eicosapentanoic, docosahexanoic fatty acids were entered as independent variables; and serum concentration of specific and total IgE antibodies as dependent variable, in a forward stepwise multivariate linear regression analysis to identify which factor(s) had the greatest influence on serum concentrations of IgE antibodies in obesity.

SECONDARY OUTCOMES:
Relationship between dietary levels of arachidonic, eicosapentanoic, docosahexanoic fatty acids and plasma concentration of leptin in obesity | one day
  Dietary intake of the omega 6 and 3 fatty acids of were analyzed in relation to plasma concentration of leptin in obese and non obese women.
Correlation between dietary arachidonic, eicosapentanoic,and docoshexanoic fatty acids and plasma concentration of adiponectin in obesity | one day
  Dietary intake of the omega 6 and 3 fatty acids of were analyzed in relation to plasma concentration of adiponectin in obese and non obese women.

REFERENCES:
- [Result] Cordain L, Eaton SB, Sebastian A, Mann N, Lindeberg S, Watkins BA, O'Keefe JH, Brand-Miller J. Origins and evolution of the Western diet: health implications for the 21st century. Am J Clin Nutr. 2005 Feb;81(2):341-54. doi: 10.1093/ajcn.81.2.341. PMID 15699220
- [Result] Linneberg A, Gislum M, Johansen N, Husemoen LL, Jorgensen T. Temporal trends of aeroallergen sensitization over twenty-five years. Clin Exp Allergy. 2007 Aug;37(8):1137-42. doi: 10.1111/j.1365-2222.2007.02760.x. PMID 17651142
- [Result] Holt PG, Macaubas C, Stumbles PA, Sly PD. The role of allergy in the development of asthma. Nature. 1999 Nov 25;402(6760 Suppl):B12-7. doi: 10.1038/35037009. PMID 10586890
- [Result] Beuther DA. Recent insight into obesity and asthma. Curr Opin Pulm Med. 2010 Jan;16(1):64-70. doi: 10.1097/MCP.0b013e3283338fa7. PMID 19844182
- [Result] Ma J, Xiao L, Knowles SB. Obesity, insulin resistance and the prevalence of atopy and asthma in US adults. Allergy. 2010 Nov;65(11):1455-63. doi: 10.1111/j.1398-9995.2010.02402.x. PMID 20456316
- [Result] Chen Y, Rennie D, Cormier Y, Dosman J. Atopy, obesity, and asthma in adults: the Humboldt study. J Agromedicine. 2009;14(2):222-7. doi: 10.1080/10599240902724051. PMID 19437281
- [Result] Husemoen LL, Glumer C, Lau C, Pisinger C, Morch LS, Linneberg A. Association of obesity and insulin resistance with asthma and aeroallergen sensitization. Allergy. 2008 May;63(5):575-82. doi: 10.1111/j.1398-9995.2007.01613.x. PMID 18394132
- [Result] Vieira VJ, Ronan AM, Windt MR, Tagliaferro AR. Elevated atopy in healthy obese women. Am J Clin Nutr. 2005 Sep;82(3):504-9. doi: 10.1093/ajcn.82.3.504. PMID 16155260
- [Result] Ouyang F, Kumar R, Pongracic J, Story RE, Liu X, Wang B, Xing H, Liu X, Li Z, Zhang W, Fang Y, Zhang S, Xu X, Wang X. Adiposity, serum lipid levels, and allergic sensitization in Chinese men and women. J Allergy Clin Immunol. 2009 Apr;123(4):940-8.e10. doi: 10.1016/j.jaci.2008.11.032. Epub 2009 Jan 9. PMID 19135238
- [Result] Kay AB. Allergy and allergic diseases. First of two parts. N Engl J Med. 2001 Jan 4;344(1):30-7. doi: 10.1056/NEJM200101043440106. No abstract available. PMID 11136958
- [Result] Wood JD, Enser M, Richardson RI, Whittington FM. Fatty acids in meat and meat products. 3rd ed. In: Chow CK ed. Fatty acids in food and health complications. Boca Raton, FL: CRC Press, 2008;87-107.
- [Result] Wortman P, Miyazaki Y, Kalupahana NS, Kim S, Hansen-Petrik M, Saxton AM, Claycombe KJ, Voy BH, Whelan J, Moustaid-Moussa N. n3 and n6 polyunsaturated fatty acids differentially modulate prostaglandin E secretion but not markers of lipogenesis in adipocytes. Nutr Metab (Lond). 2009 Jan 21;6:5. doi: 10.1186/1743-7075-6-5. PMID 19159447
- [Result] Decsi T, Molnar D, Koletzko B. Long-chain polyunsaturated fatty acids in plasma lipids of obese children. Lipids. 1996 Mar;31(3):305-11. doi: 10.1007/BF02529877. PMID 8900460
- [Result] Savva SC, Chadjigeorgiou C, Hatzis C, Kyriakakis M, Tsimbinos G, Tornaritis M, Kafatos A. Association of adipose tissue arachidonic acid content with BMI and overweight status in children from Cyprus and Crete. Br J Nutr. 2004 Apr;91(4):643-9. doi: 10.1079/BJN20031084. PMID 15035692
- [Result] Massiera F, Saint-Marc P, Seydoux J, Murata T, Kobayashi T, Narumiya S, Guesnet P, Amri EZ, Negrel R, Ailhaud G. Arachidonic acid and prostacyclin signaling promote adipose tissue development: a human health concern? J Lipid Res. 2003 Feb;44(2):271-9. doi: 10.1194/jlr.M200346-JLR200. Epub 2002 Nov 4. PMID 12576509
- [Result] Jaworski K, Ahmadian M, Duncan RE, Sarkadi-Nagy E, Varady KA, Hellerstein MK, Lee HY, Samuel VT, Shulman GI, Kim KH, de Val S, Kang C, Sul HS. AdPLA ablation increases lipolysis and prevents obesity induced by high-fat feeding or leptin deficiency. Nat Med. 2009 Feb;15(2):159-68. doi: 10.1038/nm.1904. Epub 2009 Jan 11. PMID 19136964
- [Result] Caspar-Bauguil S, Fioroni A, Galinier A, Allenbach S, Pujol MC, Salvayre R, Cartier A, Lemieux I, Richard D, Biron S, Marceau P, Casteilla L, Penicaud L, Mauriege P. Pro-inflammatory phospholipid arachidonic acid/eicosapentaenoic acid ratio of dysmetabolic severely obese women. Obes Surg. 2012 Jun;22(6):935-44. doi: 10.1007/s11695-012-0633-0. PMID 22460550
- [Result] Fain JN, Madan AK, Hiler ML, Cheema P, Bahouth SW. Comparison of the release of adipokines by adipose tissue, adipose tissue matrix, and adipocytes from visceral and subcutaneous abdominal adipose tissues of obese humans. Endocrinology. 2004 May;145(5):2273-82. doi: 10.1210/en.2003-1336. Epub 2004 Jan 15. PMID 14726444
- [Result] Snijdewint FG, Kalinski P, Wierenga EA, Bos JD, Kapsenberg ML. Prostaglandin E2 differentially modulates cytokine secretion profiles of human T helper lymphocytes. J Immunol. 1993 Jun 15;150(12):5321-9. PMID 8390534
- [Result] Bao YS, Zhang P, Xie RJ, Wang M, Wang ZY, Zhou Z, Zhai WJ, Feng SZ, Han MZ. The regulation of CD4+ T cell immune responses toward Th2 cell development by prostaglandin E2. Int Immunopharmacol. 2011 Oct;11(10):1599-605. doi: 10.1016/j.intimp.2011.05.021. Epub 2011 May 31. PMID 21635971
- [Result] Hersoug LG, Linneberg A. The link between the epidemics of obesity and allergic diseases: does obesity induce decreased immune tolerance? Allergy. 2007 Oct;62(10):1205-13. doi: 10.1111/j.1398-9995.2007.01506.x. PMID 17845592
- [Result] Couet C, Delarue J, Ritz P, Antoine JM, Lamisse F. Effect of dietary fish oil on body fat mass and basal fat oxidation in healthy adults. Int J Obes Relat Metab Disord. 1997 Aug;21(8):637-43. doi: 10.1038/sj.ijo.0800451. PMID 15481762
- [Result] Calder PC. The relationship between the fatty acid composition of immune cells and their function. Prostaglandins Leukot Essent Fatty Acids. 2008 Sep-Nov;79(3-5):101-8. doi: 10.1016/j.plefa.2008.09.016. Epub 2008 Oct 23. PMID 18951005
- [Result] Williams PB, Barnes JH, Szeinbach SL, Sullivan TJ. Analytic precision and accuracy of commercial immunoassays for specific IgE: establishing a standard. J Allergy Clin Immunol. 2000 Jun;105(6 Pt 1):1221-30. doi: 10.1067/mai.2000.105219. PMID 10856158
- [Result] Chen W, Mempel M, Schober W, Behrendt H, Ring J. Gender difference, sex hormones, and immediate type hypersensitivity reactions. Allergy. 2008 Nov;63(11):1418-27. doi: 10.1111/j.1398-9995.2008.01880.x. PMID 18925878
- [Result] Duncan MH, Singh BM, Wise PH, Carter G, Alaghband-Zadeh J. A simple measure of insulin resistance. Lancet. 1995 Jul 8;346(8967):120-1. doi: 10.1016/s0140-6736(95)92143-5. No abstract available. PMID 7603193
- [Result] Liu S, Manson JE, Stampfer MJ, Holmes MD, Hu FB, Hankinson SE, Willett WC. Dietary glycemic load assessed by food-frequency questionnaire in relation to plasma high-density-lipoprotein cholesterol and fasting plasma triacylglycerols in postmenopausal women. Am J Clin Nutr. 2001 Mar;73(3):560-6. doi: 10.1093/ajcn/73.3.560. PMID 11237932
- [Result] Black PN, Sharpe S. Dietary fat and asthma: is there a connection? Eur Respir J. 1997 Jan;10(1):6-12. doi: 10.1183/09031936.97.10010006. PMID 9032484
- [Result] Simopoulos AP. The importance of the ratio of omega-6/omega-3 essential fatty acids. Biomed Pharmacother. 2002 Oct;56(8):365-79. doi: 10.1016/s0753-3322(02)00253-6. PMID 12442909
- [Result] Daniel CR, Cross AJ, Koebnick C, Sinha R. Trends in meat consumption in the USA. Public Health Nutr. 2011 Apr;14(4):575-83. doi: 10.1017/S1368980010002077. Epub 2010 Nov 12. PMID 21070685
- [Result] Rule DC, Broughton KS, Shellito SM, Maiorano G. Comparison of muscle fatty acid profiles and cholesterol concentrations of bison, beef cattle, elk, and chicken. J Anim Sci. 2002 May;80(5):1202-11. doi: 10.2527/2002.8051202x. PMID 12019607
- [Result] Clifton PM, Condo D, Keogh JB. Long term weight maintenance after advice to consume low carbohydrate, higher protein diets--a systematic review and meta analysis. Nutr Metab Cardiovasc Dis. 2014 Mar;24(3):224-35. doi: 10.1016/j.numecd.2013.11.006. Epub 2013 Dec 20. PMID 24472635
- [Result] Melanson K, Gootman J, Myrdal A, Kline G, Rippe JM. Weight loss and total lipid profile changes in overweight women consuming beef or chicken as the primary protein source. Nutrition. 2003 May;19(5):409-14. doi: 10.1016/s0899-9007(02)01080-8. PMID 12714091
- [Result] Moreau D, Kalaboka S, Choquet M, Annesi-Maesano I. Asthma, obesity, and eating behaviors according to the diagnostic and statistical manual of mental disorders IV in a large population-based sample of adolescents. Am J Clin Nutr. 2009 May;89(5):1292-8. doi: 10.3945/ajcn.2008.26954. Epub 2009 Mar 25. PMID 19321566
- [Result] Miles EA, Aston L, Calder PC. In vitro effects of eicosanoids derived from different 20-carbon fatty acids on T helper type 1 and T helper type 2 cytokine production in human whole-blood cultures. Clin Exp Allergy. 2003 May;33(5):624-32. doi: 10.1046/j.1365-2222.2003.01637.x. PMID 12752591
- [Result] Roper RL, Brown DM, Phipps RP. Prostaglandin E2 promotes B lymphocyte Ig isotype switching to IgE. J Immunol. 1995 Jan 1;154(1):162-70. PMID 7995935
- [Result] Nagel G, Nieters A, Becker N, Linseisen J. The influence of the dietary intake of fatty acids and antioxidants on hay fever in adults. Allergy. 2003 Dec;58(12):1277-84. doi: 10.1046/j.1398-9995.2003.00296.x. PMID 14616103
- [Result] Kompauer I, Demmelmair H, Koletzko B, Bolte G, Linseisen J, Heinrich J. Association of fatty acids in serum phospholipids with hay fever, specific and total immunoglobulin E. Br J Nutr. 2005 Apr;93(4):529-35. doi: 10.1079/bjn20041387. PMID 15946416
- [Result] Krebs JD, Browning LM, McLean NK, Rothwell JL, Mishra GD, Moore CS, Jebb SA. Additive benefits of long-chain n-3 polyunsaturated fatty acids and weight-loss in the management of cardiovascular disease risk in overweight hyperinsulinaemic women. Int J Obes (Lond). 2006 Oct;30(10):1535-44. doi: 10.1038/sj.ijo.0803309. Epub 2006 Mar 21. PMID 16552404
- [Result] Tsang JY, Li D, Ho D, Peng J, Xu A, Lamb J, Chen Y, Tam PK. Novel immunomodulatory effects of adiponectin on dendritic cell functions. Int Immunopharmacol. 2011 May;11(5):604-9. doi: 10.1016/j.intimp.2010.11.009. Epub 2010 Nov 19. PMID 21094289
- [Result] De Rosa V, Procaccini C, Cali G, Pirozzi G, Fontana S, Zappacosta S, La Cava A, Matarese G. A key role of leptin in the control of regulatory T cell proliferation. Immunity. 2007 Feb;26(2):241-55. doi: 10.1016/j.immuni.2007.01.011. PMID 17307705
- [Result] Lloyd CM, Hawrylowicz CM. Regulatory T cells in asthma. Immunity. 2009 Sep 18;31(3):438-49. doi: 10.1016/j.immuni.2009.08.007. PMID 19766086
- [Result] Manigrasso MR, Ferroni P, Santilli F, Taraborelli T, Guagnano MT, Michetti N, Davi G. Association between circulating adiponectin and interleukin-10 levels in android obesity: effects of weight loss. J Clin Endocrinol Metab. 2005 Oct;90(10):5876-9. doi: 10.1210/jc.2005-0281. Epub 2005 Jul 19. PMID 16030165
- [Result] Nagel G, Koenig W, Rapp K, Wabitsch M, Zoellner I, Weiland SK. Associations of adipokines with asthma, rhinoconjunctivitis, and eczema in German schoolchildren. Pediatr Allergy Immunol. 2009 Feb;20(1):81-8. doi: 10.1111/j.1399-3038.2008.00740.x. Epub 2008 Mar 7. PMID 18331416